CLINICAL TRIAL: NCT07062211
Title: Diagnostic Accuracy of Flourodeoxyglucose-18 Positron Emission Computed Tomography in the Evaluation of Recurrent Papillary Thyroid Carcinoma With Patient's Raised Thyroglobulin Level in Lahore
Brief Title: Diagnostic Accuracy of Fluorodeoxyglucose-18 PET in the Evaluation of RPTC With Patient's Raised Thyroglobulin Level
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/908
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Papillary Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research will employ cross-sectional analytical to determine diagnostic accuracy of Flourodeoxyglucose-18 Positron Emission Computed Tomography in the evaluation of Recurrent Papillary Thyroid Carcinoma with patient's raised Thyroglobulin level in Lahore.

ELIGIBILITY:
Inclusion Criteria:

* Patients include both male and female from 18years to 80years
* Patients presented with raised thyroglobulin
* Patients with suspected diagnosis of recurrent papillary thyroid carcinoma

Exclusion Criteria:

* Patients exclude both male and female below 18years and above 80years
* All the patients presented with carcinoma other than papillary carcinoma.
* All the patients with normal thyroglobulin level.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research will employ cross-sectional analytical to determine diagnostic accuracy of Flourodeoxyglucose-18 Positron Emission Computed Tomography in the evaluation of Recurrent Papillary Thyroid Carcinoma with patient's raised Thyroglobulin level
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Nominal self admsinitered questioner | 12 Months
  Scoring in a nominal scale involves assigning a unique numerical or symbolic code to each category. For instance, in a gender survey, you might code male as "1" and female as "2." However, these codes are purely for identification and do not imply any order or magnitude

CONTACTS AND LOCATIONS:
Locations (1):
- INMOL hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No